CLINICAL TRIAL: NCT02466685
Title: Testing the Ability of JNJ(Janssen and Janssen)18038683, a Selective Serotonin (5-HT)7 Antagonist, to Improve Cognition and Reduce Residual Depressive Symptoms in Stable Bipolar Patients (18038683BCD2001)
Brief Title: Testing the Ability of JNJ-18038683 to Improve Cognition and Reduce Depressive Symptoms in Stable Bipolar Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Meltzer (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Herbert Meltzer, Professor of Psychiatry, Physiology and Pharmacology, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18038683BCD2001
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Results first posted 2023-07-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Bipolar Disorder
Keywords: Bipolar; Depression; Cognition; Cognitive
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — 3-(4-chlorophenyl)-1,4,5,6,7,8-hexahydro-1-(phenylmethyl)pyrazolo(3,4-d)azepine 2-hydroxy-1,2,3-propanetricarboxylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-18038683 (Experimental): Subjects will be randomized to receive JNJ-18038683 or placebo after the completion of the baseline assessments. Subjects randomized to JNJ-18038683 will receive 10 mg for one week, then titrate to 20 mg for the duration of the trial, with the provision for a single, downward dose adjustment for intolerance, based upon investigator judgment.
  Interventions: Drug: JNJ-18038683
- Placebo (Placebo Comparator): Placebo treatment for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-18038683 — JNJ-18038683 10-20 mg/day tablet for 8 weeks
  Arms: JNJ-18038683
Drug: Placebo — placebo tablet daily
  Arms: Placebo

SUMMARY:
The goals of this study are to evaluate the efficacy of JNJ-18038683 in an 8 week trial to ameliorate the cognitive deficit and reduce residual depressive symptoms in 60 stable bipolar outpatients receiving treatment for depression. JNJ-18038683 will be studied and compared with placebo as adjunctive treatment to standard pharmacologic treatment for bipolar disorder.

DETAILED DESCRIPTION:
Most, but not all, patients with bipolar disorder (BPD) have clinically significant cognitive impairment. Impairment is present in both the manic and depressed phases of BPD, as well as in euthymic periods. The percentage of BPD patients with cognitive impairment (CIBD) varies among studies, with 40-60% representing the best estimate. The weight of the evidence supports no overall difference in the type and severity of cognitive impairment in any phase of BPD, i.e. it is a stable trait feature of BPD, albeit variable from one patient to another. The most commonly affected cognitive domains are speed of processing, declarative memory, attention and working memory. Although CIBD is milder in severity than the cognitive impairment associated with schizophrenia (CIAS), on average, as in schizophrenia, CIBD has a major impact on function and quality of life in most patients, particularly because the greater preservation of function of BPD enables them to engage in activities which are more dependent on intact cognitive function. Thus, it is highly likely that improvement in CIBD will have valuable clinical benefit, especially with regard to quality of life measures. It is reasonable to predict that treatments effective to improve CIBD could also be beneficial for CIAS. Efficacy for cognitive impairment is likely to be greater in BPD than schizophrenia, because the baseline severity is milder in the former. Despite this strong rationale for targeting CIBD, there has been minimal focus on clinical trials to improve CIBD, perhaps because so many resources have been devoted to the effort to treat CIAS, but lack of appreciation of the severity of CIBD and its importance as a determinant of functional outcome in BPD may be the most important factors.

In a recent study of CIBD, using the MATRICS Consensus Cognitive Battery (MCCB), impairment was found in both treatment resistant BP I and II depressed inpatients within all MCCB domains. The greatest impairment was evident in speed of processing, declarative memory and attention. The impairment was numerically greater in BP I than BP II patients but the difference was not significant. Compared to normal controls, the deficits, in BP 1 patients, in speed of processing was 1.2SD, in attention, 1.0 SD, and in verbal learning, 1.8 SD. The least affected domain was visual learning, with a mean deficit of 0.8SD compared to normal controls. The mean composite score deficit was 1.25 SD. Medication for BPD, particularly mood stabilizers, may adversely affect some domains of cognition in BPD. However, antidepressant medications have not been found to affect the severity of cognitive impairment in major depression or BPD.

Based on the pre-clinical, pro-cognitive effects of 5-HT7 antagonism in our laboratory, along with the reported pre-clinical antidepressant effects of JNJ-18038683, we propose to conduct a randomized, placebo- controlled parallel, design study to assess the effects of JNJ-18038683 on multiple domains of cognition and mood symptoms. Since our preclinical studies show that 5-HT7 receptor blockade is highly effective in improving declarative memory in rodents, the declarative memory measures will be the primary outcome measures.

Due to the effect of JNJ-18038683 on depressive symptoms in preclinical paradigms, we will investigate the following in the clinical trial the potential antidepressant effect of JNJ-18038683 on patients with baseline MADRS score between 8 and 20.

ELIGIBILITY:
Inclusion Criteria

1. All participants must have signed an informed consent document indicating they understand the purpose of the study and the procedures required for the study and are willing to participate by complying with the study procedures and restrictions.
2. Male or female individuals of any race; between 18 to 60 years of age, inclusive.
3. Resides in a stable living situation, according to the investigator's judgment.
4. Diagnosis of bipolar disorder I or II for at least 1 year in duration, as established by the SCID-I, and verified with medical records and/or confirmation of diagnosis by treating clinician. Patients will be in a nonacute phase at the time of initial screening and have been so for at least 1 month.
5. No more than moderate clinical symptom burden severity, as defined by the following: Montgomery Asberg Depression Rating Scale < 20 Young Mania Rating Scale <12
6. Individuals medically stable enough to complete an 8 week clinical trial, in the judgment of the investigator
7. Women of childbearing potential must have a negative pregnancy serum test at screening, negative pregnancy urine test at baseline, and agree to use adequate protection (i.e. double barrier method) for birth control.
8. Antidepressant (AD) medications are allowed if the subject has been treated with a stable dose for at least 2 months before screening.
9. Individuals receiving a single mood stabilizer (e.g., lithium. valproate, or lamictal) are allowed if a stable dose has been maintained for at least 2 months prior to screening.
10. Individuals may be receiving one treatment of each the following groups:

    antidepressants, mood stabilizers, and atypical antipsychotics other than clozapine, but not more than one from each group.
11. Individuals taking ripseridone, lurasidone, or ziprasidone must be currently taking < doses of 3mg, 40mg, and, 80mg, respectively.
12. Subjects may be treated with inclusionary antipsychotic drugs as long as they are on a stable dose of injectable medication for 2 months or a sable dose of an oral medication for 1 month. Exclusionary antipsychotic drugs are listed in Appendix 2 in the protocol.
13. Patients with a history of compliance with a drug treatment regimen for bipolar disorder, as noted in medical/psychiatric history.
14. CNS stimulants (e.g., Adderall, Ritalin) are permitted if the participant is stable on their dosage of medication for 1 month before screening and cannot change dosage throughout the study.
15. Able to complete cognition assessments in English
16. Individuals must demonstrate a substantive cognitive deficit, as measured by the Trails A, Hopkins Verbal Learning Test (HVLT), and the Letter Number Span, administered at the screening visit. Eligible individuals will have an established cognitive deficit as measured by one or more of these tests, scoring below the 75th percentile, using comparative norms according to age, gender, and education.
17. Able to understand and complete cognition assessments

Exclusion Criteria

1. Failure to perform screening or baseline examinations
2. Hospitalization within 8 weeks before screening, or change in mood stabilizing or antidepressant medication or dose within 2 months prior to screening.
3. Individuals who have participated in another clinical study within the past 2 months.
4. Individuals with tardive dyskinesia.
5. Individuals with other DSM-V Axis I or Axis II primary diagnoses.
6. Diagnosis of alcohol or substance use disorder within the past 3 months.
7. Subject assessed to be at significant suicide risk based on responses to the Columbia Suicide Severity Rating Scale (C-SSRS).
8. History of myocardial infarction, unstable angina, uncontrolled hypotension or hypertension within 3 months before screening.
9. Clinically significant abnormality on screening ECG.
10. Alanine transaminase (ALT) or aspartate transaminase (AST) > 2.5 times the upper limit of normal (ULN).
11. History of stroke, brain tumor, head trauma with loss of consciousness, or other clinically significant neurological condition within 12 months before screening.
12. Individuals with other uncontrolled medical conditions, in the opinion of the investigator.
13. Use of drugs known to be metabolized by CYP2D6.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2021-09 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine; Department of Psychiatry and Behavioral Sciences, Chicago, Illinois, United States

REFERENCES:
- [Derived] Arshadi M, Elmaadawi AZ, Nasr S, Jayathilake K, Rassnick S, Ford L, Drevets WC, Meltzer HY. Lack of Efficacy of JNJ-18038683 on Cognitive Impairment in Patients With Stable Bipolar Disorder. J Clin Psychopharmacol. 2024 Sep-Oct 01;44(5):481-491. doi: 10.1097/JCP.0000000000001889. PMID 39250138

RESULTS

PARTICIPANT FLOW:
Groups:
- JNJ-18038683: Subjects will be randomized to receive JNJ-18038683 or placebo after the completion of the baseline assessments. Subjects randomized to JNJ-18038683 will receive 10 mg for one week, then titrate to 20 mg for the duration of the trial, with the provision for a single, downward dose adjustment for intolerance, based upon investigator judgment.
  JNJ-18038683: JNJ-18038683 10-20 mg/day for 8 weeks
- Placebo: Placebo treatment for 8 weeks.
  JNJ-18038683: JNJ-18038683 10-20 mg/day for 8 weeks
Period: Overall Study
Arm/Group | JNJ-18038683 | Placebo
Started | 30 | 30
Completed | 22 | 26
Not Completed | 8 | 4
Not completed — Adverse Event | 5 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JNJ-18038683 | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (12.1) | 37.4 (11.0) | 38.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 8 | 14 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 10 | 15
  White | 22 | 19 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Verbal Fluency [Least Squares Mean (Standard Deviation); unit: units on a scale] — Verbal Fluency, as a primary outcome measure, is one of the Cognitive battery tests used to evaluate neurocognitive functions, i.e: speed of processing, attention/vigilance, working memory, verbal learning, visual learning. Higher schore means better outcome
  units on a scale | 35.87 (2.12) | 40.07 (2.16) | 38.82 (2.14)

OUTCOME MEASURES:

1. Primary Outcome: The 8-week Evaluation of Verbal Fluency Performance After Randomization
Description: Change in a score of Verbal Fluency from baseline to week 8 A higher amount of change represents a better outcome V.F., as a primary outcome measure, is one of the Cognitive battery tests used to evaluate neurocognitive functions, i.e., speed of processing, attention/vigilance, working memory, verbal learning, and visual learning.
  The way to calculate the score: the participant is asked to produce as many words as possible from a category in a given time and each correct word gets 1 score Min raw score:0 Max raw score:60
Time Frame: Baseline and week 8
Population: Although the total number of participants in each group was 30, the analysis was only done for those who had completed all study visits.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- JNJ-18038683: JNJ-18038683: JNJ-18038683 10-20 mg/day for 8 weeks
Arm/Group | JNJ-18038683 | Placebo
Number analyzed (Participants) | 22 | 26
score on a scale | 39.44 (1.31) | 41.12 (1.33)
Statistical Analysis 1: Comparison: JNJ-18038683 vs Placebo; Test type: Superiority; p < 0.05, ANCOVA; Mean Difference (Final Values) = 5, Standard Deviation 9.4

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Secondary outcome measures will include mean changes of the Montgomery-Asberg Depression Rating Scale (MADRS) total score from baseline to week 8.
  The MADRS will be utilized to assess a subject's level of depressive symptoms and must be administered using a structured interview guide.
  This scale consists of 10 items, each with seven defined grades of severity (zero to six), and min score of 0, and a max score of 60.
  Higher values represent a worse outcome. Notably, mean changes were not statistically significant in both groups.
Time Frame: Baseline to week 8
Population: Although the total number of each group was 30, only data of the participants who completed week eight were analyzed on MADRS.
  ANCOVA analysis for comparing the result of the Montgomery Asberg Depression rating scale between JNJ-18038683 and the placebo group, based on the least-square means and standard errors, will be the statistical method. The Missing data will be imputed by MMRM.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Participants Receiving JNJ-18038683 Tablet From Baseline to week8: Subjects who were randomized to JNJ-18038683 and completed baseline and week eight visits were eligible participants of this group. Subjects received 10 mg for one week, then titrated to 20 mg for the duration of the trial.
  ANCOVA analysis for comparing the result of the Montgomery Asberg Depression rating scale between JNJ-18038683 and the placebo group, based on the least-square means and standard Errors.
Arm/Group | Participants Receiving JNJ-18038683 Tablet From Baseline to week8 | Placebo
Number analyzed (Participants) | 22 | 26
score on a scale
  MADRS baseline score | 2.93 (0.71) | 3.37 (0.71)
  MADRS week 8 score | 6.63 (1.26) | 5.89 (1.26)

3. Secondary Outcome: Clinical Global Impression Severity of the Subject With Bipolar Disorder Scale( CGI-S in BP) Change From Baseline to Week 8
Description: We assessed the clinical global Impression severity (CGI-S) scores change in JNJ-18038683 and the placebo group as an additional endpoint.
  The scale rates the subject's Severity of Illness (CGI-BPSeverity: mania, depression, and overall bipolar illness). Using ANCOVA analysis to assess changes from baseline to week 8, based on the least-square means and standard errors was the method.
  CGI-S scores range from 0 to 7. Higher scores mean a worse outcome.
Time Frame: Baseline to 8 weeks
Population: Although the total number of participants in each group was 30, the analysis was only done for those who had completed all study visits. Using ANCOVA analysis to assess changes from baseline to week 8, based on the least-square means and standard errors was the method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- JNJ-18038683: Subjects randomized to JNJ-18038683 will receive 10 mg for one week, then titrate to 20 mg for the duration of the trial, with the provision for a single, downward dose adjustment for intolerance, based upon investigator judgment. Only participants who completed the baseline and week 8 visit are eligible for this measure.
Arm/Group | JNJ-18038683 | Placebo
Number analyzed (Participants) | 22 | 26
score on a scale
  CGI-S baseline score | 2.78 (0.19) | 2.63 (0.19)
  CGI-S week 8 score | 2.59 (0.19) | 2.37 (0.19)

ADVERSE EVENTS:
Time Frame: During the study, from baseline to week12 (from baseline to 4 weeks after the study completion)
Description: The total number affected by any Serious Adverse Event was 4 patients but 5 events.
  Regarding Non-Serious Adverse Events, reports are according to the threshold of 5%
Arm/Group | JNJ-18038683 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/30 | 1/30
Other Adverse Events (participants affected / at risk) | 6/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JNJ-18038683 (N=30) | Placebo (N=30)
Serious Adverse Event (Psychiatric disorders) | 2 (3) | 1 (1) — Suicidal ideation in 2 patients in JNJ-18038683 and 1 patient in the Placebo group
Serious Adverse events (Gastrointestinal disorders) | 1 (1) | 0 (0) — Abdominal pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JNJ-18038683 (N=30) | Placebo (N=30)
Non-Serious Adverse Events (Psychiatric disorders) | 6 (7) | 0 (0) — Sleep disorder
Non-Serious Adverse Events (Gastrointestinal disorders) | 0 (0) | 2 (5) — Nausea
Non-Serious Adverse Events (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Upper respiratory infection
Non-Seriuos Adverse event (Psychiatric disorders) | 0 (0) | 2 (2) — Mood lability
Non-Serious Adverse Events (General disorders) | 3 (3) | 0 (0) — Dizziness
Non-Serious Adverse Events (General disorders) | 2 (2) | 0 (0) — Dehydration
Non-Serious Adverse Events (Psychiatric disorders) | 3 (3) | 0 (0) — Exessive sleepiness
Non-Serious Adverse Events (Psychiatric disorders) | 2 (2) | 0 (0) — Restlessness
Non-Serious Adverse Events (Ear and labyrinth disorders) | 2 (2) | 0 (0) — Ear ringing
Non-Serious Adverse Events (Nervous system disorders) | 2 (5) | 5 (5) — Headache
Non-Serious Adverse Events (Gastrointestinal disorders) | 2 (2) | 0 (0) — Stomach pain
Non-Serious Adverse Events (Gastrointestinal disorders) | 2 (3) | 0 (0) — Heartburn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT02466685/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT02466685/SAP_001.pdf
  • Informed Consent Form (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/85/NCT02466685/ICF_002.pdf